CLINICAL TRIAL: NCT05395988
Title: Hand Hygiene of Kindergarten Children: Understanding the Effect of Live Feedback on Hand Washing Behavior, Self-Efficacy and Motivation of Young Children
Brief Title: Hand Hygiene of Kindergarten Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Otto-Friedrich-University Bamberg (Other)
Collaborators: University of Turku (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: Hand hygiene kindergarten
Record Dates: First submitted 2022-03-25; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Hand Hygiene; Hand Washing

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (No Intervention): The control group receives no screen next to the sink.
- Instruction group (Experimental): The reward group receives a screen next to each sink in kindergarten. On the screen, hand washing instructions are shown during hand washing. After a defined time period, the screen is removed.
  Interventions: Device: Digital hand washing instructions
- Reward group (Experimental): The reward group receives a screen next to each sink in kindergarten. On the screen, hand washing instructions are shown during hand washing. If hands are washed correctly (time and soap usage), a reward (animal animation) is shown on the screen.
  After a defined time period, the screen is removed.
  Interventions: Device: Digital hand washing reward
- Reward plus instruction-only group (Experimental): The reward plus instruction group receives a screen next to each sink in kindergarten.
  On the screen, hand washing instructions are shown during hand washing. If hands are washed correctly (time and soap usage), a reward (animal animation) is shown on the screen.
  After a defined time period, the screen only shows instructions, the reward is not shown anymore.
  After a defined time period, the screen is removed.
  Interventions: Device: Digital hand washing instructions; Device: Digital hand washing reward

INTERVENTIONS:
Device: Digital hand washing instructions — Tablet displaying animated hand washing instructions
  Arms: Instruction group; Reward plus instruction-only group
Device: Digital hand washing reward — Tablet displaying animated hand washing instructions and animated animals as reward
  Arms: Reward group; Reward plus instruction-only group

SUMMARY:
Randomized controlled trial to further assess the impact of a digital intervention on hand hygiene of young children. Children in intervention kindergartens will see live instructions and feedback on their hand washing activity in reals-time / while washing hands. Aim of the study is to better understand behavior change of young children.

ELIGIBILITY:
Inclusion Criteria:

* children attending kindergarten

Exclusion Criteria:

* none

Ages: 2 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2022-10 (Estimated); Study Completion 2022-10 (Estimated)

PRIMARY OUTCOMES:
Handwashing motivation of children (measured as soaping time by digital system). | up to 3 months
  Motivation of children, measured as soaping time (activity level) by digital system. Activity level is used as a proxy for motivation.
Handwashing motivation of children (investigated with observation questionnaire for children in kindergarten) | up to 3 months
  Motivation of children, investigated with observation questionnaire (covering different steps of handwashing) of children while washing hands in kindergarten. In the observation questionnaire, each step of handwashing is rated on a scale (with highest number meaning highest compliance to handwashing instructions). Activity level (as measured by observation questionnaire) is used as a proxy for motivation.
Self-efficacy of children (investigated with interviews with children) | up to 3 months
  Self-efficacy of children is measured in interviews with the children. The interview questionnaires for the children are based on Bandura's concept of self-efficacy. The scale that is used in the interview questionnaires is specially developed for our experiment.
Self-efficacy of children (investigated with interviews with staff) | up to 3 months
  Self-efficacy of children is measured in interviews with the kindergarten staff. The interview questionnaires for the staff (for evaluating children's self-efficacy) are based on Bandura's concept of self-efficacy. The scale that is used in the interview questionnaires is specially developed for our experiment.

SECONDARY OUTCOMES:
Sickness days of children (as recorded by kindergarten management) | Up to one year
  Sickness days of children, recorded by kindergarten management on a daily basis.

CONTACTS AND LOCATIONS:
Overall Officials: Sanna Salanterä, Prof. Dr., Principal Investigator — University of Turku; Joanna Graichen, M.Sc., Principal Investigator — Otto-Friedrich-University Bamberg; Anni Pakarinen, PhD, Principal Investigator — University of Turku; Carlo Stingl, M.Sc., Principal Investigator — Otto-Friedrich-University Bamberg; Riitta Mieronkoski, Principal Investigator — University of Turku; Glenda Dangis, Principal Investigator — University of Turku
Locations (2):
- University of Turku, Turku, Finland
- Otto-Friedrich-University Bamberg, Bamberg, Germany

REFERENCES:
- [Derived] Dangis G, Terho K, Graichen J, Gunther SA, Rosio R, Salantera S, Staake T, Stingl C, Pakarinen A. Hand hygiene of kindergarten children-Understanding the effect of live feedback on handwashing behaviour, self-efficacy, and motivation of young children: Protocol for a multi-arm cluster randomized controlled trial. PLoS One. 2023 Jan 24;18(1):e0280686. doi: 10.1371/journal.pone.0280686. eCollection 2023. PMID 36693062